CLINICAL TRIAL: NCT01399489
Title: The Effect of Short-term Aerobic Training on Arterial Stiffness and Blood in Chronic Kidney Disease (CKD) Patients
Brief Title: Aerobic Training and Arterial Stiffness in Chronic Kidney Disease (CKD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Springfield College (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samuel A. Headley, Professor , Exercise Science, Springfield College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R15HL096097-01 (NIH)
Record Dates: First submitted 2011-01-31; First posted 2011-07-21 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Kidney Disease; Hypertension; Diabetes
Keywords: Aerobic exercise; Moderate intensity; Ambulatory blood pressure; Post exercise hypotension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Diabetes Mellitus; Post-Exercise Hypotension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): Individuals randomized to this arm get 48 sessions of personal training in a state of the art fitness facility
  Interventions: Behavioral: Exercise training
- Control (No Intervention): Individuals in the control arm are expected to continue to live normally, following their doctor's advice but not engage in any formal exercise training.

INTERVENTIONS:
Behavioral: Exercise training — Participants receive 16 weeks of moderate intensity aerobic training under the supervision of personal trainers. Each session lasts from 15 to 55 minutes depending upon patient tolerance
  Other Names: Non-pharmacologic; Lifestyle
  Arms: Exercise training

SUMMARY:
The current study is designed to examine the impact of 16 weeks of moderate intensity aerobic training on arterial stiffness and blood pressure in stage 3 chronic kidney disease (CKD) patients. The investigators hypothesize that short term aerobic training will improve the stiffness of arteries in CKD patients.

DETAILED DESCRIPTION:
The focus of the current research group is to examine the impact of lifestyle interventions on the development of cardiovascular disease (CV) in chronic kidney disease (CKD) patients. The study being proposed is to determine the effect of short-term aerobic training on arterial stiffness and blood pressure (BP) in CKD patients. Arterial stiffness has been chosen as a dependent variable since it is one of the most important predictors of CV complications while hypertension is known to play a critical role both in the development of CV and in the progression of CKD (6, 41). The specific aims of the study are: (a) to determine the effect of short-term aerobic training on arterial stiffness in CKD patients, (b) to determine the effect of short-term aerobic training on resting and ambulatory blood pressures (ABP) in CKD patients and (c) to determine the effect of short-term aerobic training on the acute post-exercise blood pressure response in CKD patients since acute responses may be related to changes following a period of chronic training. Fifty, 35-70 yr old, stage 3 CKD patients, with either diabetes or hypertension as the primary cause of their CKD will be recruited for this study. Subjects will be randomly assigned to either the exercise group (ExG = 25) or to the control group (CG = 25). At the start of the study each subject will attend 4 research sessions. During the first session, resting and 24 hr ABP readings will be recorded. In the second session, anthropometric measures, peak oxygen uptake (VO2peak), and ABP values will be measured. Sessions 3 & 4 will be performed in random order. During these sessions, pulse wave velocity (PWV), augmentation index (AIx) and BP will be measured at baseline after a rest period. Subjects will then either walk for 30 min at 50-60% of VO2 peak, or sit quietly for an equal period of time. BP will be monitored for 60 min in recovery following exercise and ABP will be taken during the subsequent 24 hrs. ExG will perform supervised aerobic training for 45-50 min, 3 times per week, at a moderate intensity, for 16 weeks. CG will continue their activities of daily living but will not be given an exercise program. All subjects will be retested at week 8 for BP, ABP, and arterial stiffness and at week 16 for all variables. After 16 weeks of the study both groups will be retested using identical procedures as at baseline. A series of 2 X 2 analyses of covariance with age, baseline PWV, AIx and BP as the covariates, will be used to determine the effect of the 16 week intervention period on the primary outcome variables. A 2 X 7 X 2, mixed factorial repeated measures ANOVA will be used to analyze the post-exercise data while a Pearson Moment Correlation Coefficient will be computed to examine the relationship between post-exercise acute responses and BP changes following chronic training. An alpha level of 0.05 will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 Chronic Kidney Disease (CKD)
* Primary diagnosis hypertension or diabetes

Exclusion Criteria:

* Smokers
* Individuals < 35 or > 70 years of age
* Any contraindicators to exercise training as defined by the ACSM guidelines (GETP8)

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Arterial stiffness (pulse wave velocity) | Change from Baseline in PWV at 16 weeks
  Arterial stiffness is measured via pulse wave velocity. In addition augmentation index is also being assessed. Blood pressure is being measured under resting conditions and via 24 hr ambulatory devices.

SECONDARY OUTCOMES:
Change in Resting blood pressure from Baseline | Baseline prior to acute exercise vs post acute exercise
  Resting blood pressure is measured at baseline before an acute bout of exercise and for 1 hour in the laboratory after 40 min of exercise. This is repeated after 16 weeks of training or after the 16 control period
Change in Resting blood pressure after 16 weeks of training | Change in resting blood pressure from baseline at 16 weeks of training
  Resting blood pressure is measured at baseline before an acute bout of exercise and for 1 hour in the laboratory after 40 min of exercise. This is repeated after 16 weeks of training or after the 16 control period

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Headley, Ph.D, Principal Investigator — Sprtingfield College
Locations (1):
- Athletic Training and Exercise Science Building, Springfield, Massachusetts, United States